CLINICAL TRIAL: NCT04440150
Title: Preoperative Immature Granulocyte Count and Percentage for Complicated and Uncomplicated Appendisitis
Brief Title: Preoperative Immature Granulocyte Count and Percentage for Acute Appendisitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Mehmet Buğra Bozan, Professor, Assistant, Kahramanmaras Sutcu Imam University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 180
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Acute Appendicitis
Keywords: Acute Appendicitis; Complicated Acute Appandicitis; Emergent Surgery; Immature Granulocyte Count; Immature Granulocyte Percentage
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Intervention Model Description: Retrospective Cohort Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complicated Acute Appendicitis (Other): The patients were assigned to the complicated acute appendicitis group (Group C) based on the preoperative imaging findings (periappendiceal abscess formation or significant periappendiceal fat tissue contamination in ultrasonography and computed tomography), intraoperative exploration findings (presence of gangrenous appendicitis, perforation or abscess formation), and pathological examination findings (acute phlegmonous appendicitis, acute gangrenous appendicitis or acute perforated appendicitis).
  Interventions: Procedure: Appendectomy
- Uncomplicated Acute Appendicitis (Other): The patients were assigned to the uncomplicated acute appendicitis group (Group UC) based on the increased diameter and wall thickness of the appendix and detection of minimal contamination in the surrounding fat tissue in the imaging tests; the presence of edema and the absence of gangrene, perforation or abscess in the the exploratory surgery of appendix, and confirmation of the diagnosis of acute appendicitis by the pathological examination findings
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Procedure: Appendectomy — Open or Laparascopic Surgery

SUMMARY:
Appendectomy is the most effective treatment option for acute appendisitis, which is the most commen emergent surgical pathology. However with in time period, surgical treatment borders are narrowed. Especially in uncomplicated acute appendicitis cases, nonoperative management (NOM) with antibiotherapies becomes primary treatment option. The COVID-19 pandemic, which is caused by 2019 novel coronavirus (2019-nCoV) and we encountered in the current process, has led to the re-questioning of surgical elective and emergency cases. Serious complications and increased mortality rates of the 2019-nCoV creates a novel problems of patient selection for emergent surgery and health care workers faced with potential health problems. As the same as the other surgical procedures, in the uncomplicated acute appendisitis cases NOM become more mandantory. NOM of uncomplicated acute appendisitis doen't increase perforation risk and general practice for decreasing surgical complications in the COVID-19 pandemic period. Additionally complicated acute appendicitis accounts for 20 to 30% of the patients undergoing appendectomy and lead to increased risk of postoperative complications, delayed recovery and longer hospital stay. Therefore, early diagnosis of complicated acute appendicitis is important; however, the most appropriate and inexpensive diagnostic method to make this diagnosis has not been established yet. Although the use of imaging methods is widespread, these methods are not accessible in many rural hospitals due to the high costs and unavailability of specialists. Thus, the need for an inexpensive and effective diagnostic technique allowing to make a differential diagnosis has not been met yet. For this purpose, several inexpensive and easily accessible blood parameter tests have been proposed; including the white blood cell count, immature granulocyte (IG) percentage, C-reactive protein levels or the neutrophil-to-lymphocyte ratio.

An increase in the IG count shows that the bone marrow is active. This parameter has been used as a prognostic factor in many infectious and non infectious diseases including sepsis, acute pancreatitis, and acute myocardial infarction. The Immature granulocyte (IG) fraction includes promyelocytes, myelocytes, and metamyelocytes but not band neutrophils or myeloblasts. The IG count and percentage has become an easy-to-use method, especially with the introduction of technological advances, as it can be easily determined using the results of a routine complete blood count.

It is aimed to efficacy of IG count and percentage which are calculated automatically in CBC samples, to differatiate the complicated and uncomplicated acute appendicitis cases with a cheap, easily applicable and cost effective test, especially in rural areas without enough diagnostic tests in COVID-19 pandemy.

DETAILED DESCRIPTION:
The data of 146 patients elder than 18 years, who admitted to the Emergency Department and General Surgery outpatient clinic with the complaint of abdominal pain diagnosed with acute appendicitis and who were operated by the same surgical team between June 2018 and June 2019 were evaluated retrospectively after the approval of the local ethics committee. Patients' data were obtained by reviewing the patient follow charts, laboratory findings in the the electronic database of the hospital and epicrisis forms. Totally 76 patients excluded from the study; 22 patients were excluded because of the pathological diagnosis did not confirm acute appendicitis (negative appendectomies and appendiceal mucinous cystadenomas), 54 patients who were operated by the other surgical team were excluded.

The patients were assigned to the complicated acute appendicitis group (Group C) based on the preoperative imaging findings (periappendiceal abscess formation or significant periappendiceal fat tissue contamination in ultrasonography and computed tomography), intraoperative exploration findings (presence of gangrenous appendicitis, perforation or abscess formation), and pathological examination findings (acute phlegmonous appendicitis, acute gangrenous appendicitis or acute perforated appendicitis). The patients were assigned to the uncomplicated acute appendicitis group (Group UC) based on the increased diameter and wall thickness of the appendix and detection of minimal contamination in the surrounding fat tissue in the imaging tests; the presence of edema and the absence of gangrene, perforation or abscess in the the exploratory surgery of appendix, and confirmation of the diagnosis of acute appendicitis by the pathological examination findings [17-20].

The WBC, IG count and IG percentage automatically calculated in the complete blood count (CBC) parameters. WBC count, neutrophil count, lymphocyte count, and IG% were measured using an automated hematological analyzer (XN 3000; Sysmex Corp., Kobe, Japan) from blood samples obtained at the initial admission to the emergency department . Neutrophyl and Lymphocyte counts were obtained from automatically from the CBC parameters and NLR was calculated manually.

The demographic data (age, sex) of the patients, the white blood cell count (WBC), the neutrophil-to-lymphocyte ratio (NLR), and the IG count and percentage were evaluated retrospectively.

Statistical Analysis Statistical analyses were performed with the IBM Statistical Package for Social Sciences (SPSS) version 20.0 software. The student t-test or Mann-Whitney U test were used for analyzing the quantitive values based on normality of the distrubution calculated with Shapiro Wilk Test. The chi-square test or Fischer's exact test was used for analyzing the categorical data. ROC analysis was used to determeine spesivity and sensitivity of the parameters. Binary logistic regression analysis was performed to determine the preoperative diagnostic accuracy of the parameters. The quantitive data were given mean ± standard deviation (minimum - maximum values) or median (minimum - maximum values). The qualitative values were given number of cases (n) and percentage (%). A p-value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years,
* Patients diagnosed as acute appenditicitis cases according to clinical (preoperative and peroperative) and preoperative laboratory findings and imaging modalities (ultrasound, computed tomography), and pathologic results
* Patients who were operated by the same surgical team of the Kahramanmaras Sutcu Imam University Hospital.

Exclusion Criteria:

* Patients younger than 18 years,
* Negative appendectomies according to peroperative findings and pathologic findins
* Patients whose data were not available
* Patients who were operated by the other surgical team of the Kahramanmaras Sutcu Imam University.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Preoperative IG count of the patients to differentiate complicated and uncomplciated acute appendicitis | Preoperative
  Preoperative IG count of the patients to differentiate complicated and uncomplciated acute appendicitis
Preoperative IG count for selection of medical treatment patients of noncomplicated acute appendicitis | Preoperative
  Preoperative IG count of the patients to select medically treatment patients of noncomplicated acute appendicitis
Preoperative IG percentage of the patients to differentiate complicated and uncomplciated acute appendicitis | Preoperative
  Preoperative IG percentage of the patients to differentiate complicated and uncomplciated acute appendicitis
Preoperative IG percentage for selection of medical treatment patients of noncomplicated acute appendicitis | Preoperative
  Preoperative IG percentage of the patients to select medically treatment patients of noncomplicated acute appendicitis

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü İmam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kirkil C, Yigit MV, Aygen E. Long-term results of nonoperative treatment for uncomplicated acute appendicitis. Turk J Gastroenterol. 2014 Aug;25(4):393-7. doi: 10.5152/tjg.2014.7192. PMID 25254521
- [Background] Gok AFK, Eryilmaz M, Ozmen MM, Alimoglu O, Ertekin C, Kurtoglu MH. Recommendations for Trauma and Emergency General Surgery Practice During COVID-19 Pandemic. Ulus Travma Acil Cerrahi Derg. 2020 Apr;26(3):335-342. doi: 10.14744/tjtes.2020.79954. PMID 32394416
- [Background] Hogan A. COVID-19 and emergency surgery. Br J Surg. 2020 Jun;107(7):e180. doi: 10.1002/bjs.11640. Epub 2020 Apr 24. No abstract available. PMID 32329524
- [Background] De Simone B, Chouillard E, Di Saverio S, Pagani L, Sartelli M, Biffl WL, Coccolini F, Pieri A, Khan M, Borzellino G, Campanile FC, Ansaloni L, Catena F. Emergency surgery during the COVID-19 pandemic: what you need to know for practice. Ann R Coll Surg Engl. 2020 May;102(5):323-332. doi: 10.1308/rcsann.2020.0097. Epub 2020 Apr 30. PMID 32352836
- [Background] Collard M, Lakkis Z, Loriau J, Mege D, Sabbagh C, Lefevre JH, Maggiori L. Antibiotics alone as an alternative to appendectomy for uncomplicated acute appendicitis in adults: Changes in treatment modalities related to the COVID-19 health crisis. J Visc Surg. 2020 Jun;157(3S1):S33-S42. doi: 10.1016/j.jviscsurg.2020.04.014. Epub 2020 Apr 24. PMID 32362368
- [Background] Kelly ME, Murphy E, Bolger JC, Cahill RA. COVID-19 and the treatment of acute appendicitis in Ireland: a new era or short-term pivot? Colorectal Dis. 2020 Jun;22(6):648-649. doi: 10.1111/codi.15141. Epub 2020 May 31. No abstract available. PMID 32403188
- [Background] Diaz-Barrientos CZ, Aquino-Gonzalez A, Heredia-Montano M, Navarro-Tovar F, Pineda-Espinosa MA, Espinosa de Santillana IA. The RIPASA score for the diagnosis of acute appendicitis: A comparison with the modified Alvarado score. Rev Gastroenterol Mex (Engl Ed). 2018 Apr-Jun;83(2):112-116. doi: 10.1016/j.rgmx.2017.06.002. Epub 2018 Feb 6. English, Spanish. PMID 29426650
- [Background] Park JS, Kim JS, Kim YJ, Kim WY. Utility of the immature granulocyte percentage for diagnosing acute appendicitis among clinically suspected appendicitis in adult. J Clin Lab Anal. 2018 Sep;32(7):e22458. doi: 10.1002/jcla.22458. Epub 2018 Apr 30. PMID 29708633
- [Background] Khan MS, Siddiqui MTH, Shahzad N, Haider A, Chaudhry MBH, Alvi R. Factors Associated with Complicated Appendicitis: View from a Low-middle Income Country. Cureus. 2019 May 28;11(5):e4765. doi: 10.7759/cureus.4765. PMID 31363446
- [Background] Hakkoymaz H, Nazik S, Seyithanoglu M, Guler O, Sahin AR, Cengiz E, Yazar FM. The value of ischemia-modified albumin and oxidative stress markers in the diagnosis of acute appendicitis in adults. Am J Emerg Med. 2019 Nov;37(11):2097-2101. doi: 10.1016/j.ajem.2019.03.005. Epub 2019 Mar 7. PMID 30871739
- [Background] Yazar FM, Urfalioglu A, Bakacak M, Boran OF, Bulbuloglu E. Efficacy of the Evaluation of Inflammatory Markers for the Reduction of Negative Appendectomy Rates. Indian J Surg. 2018 Feb;80(1):61-67. doi: 10.1007/s12262-016-1558-y. Epub 2016 Oct 18. PMID 29581687
- [Background] van der Geest PJ, Mohseni M, Brouwer R, van der Hoven B, Steyerberg EW, Groeneveld AB. Immature granulocytes predict microbial infection and its adverse sequelae in the intensive care unit. J Crit Care. 2014 Aug;29(4):523-7. doi: 10.1016/j.jcrc.2014.03.033. Epub 2014 Apr 5. PMID 24798344
- [Background] Sauneuf B, Bouffard C, Cornet E, Daubin C, Desmeulles I, Masson R, Seguin A, Valette X, Terzi N, Parienti JJ, du Cheyron D. Immature/total granulocyte ratio: a promising tool to assess the severity and the outcome of post-cardiac arrest syndrome. Resuscitation. 2014 Aug;85(8):1115-9. doi: 10.1016/j.resuscitation.2014.04.017. Epub 2014 Apr 30. PMID 24795281
- [Background] Unal Y. A new and early marker in the diagnosis of acute complicated appendicitis: immature granulocytes. Ulus Travma Acil Cerrahi Derg. 2018 Sep;24(5):434-439. doi: 10.5505/tjtes.2018.91661. PMID 30394497
- [Background] Ayres LS, Sgnaolin V, Munhoz TP. Immature granulocytes index as early marker of sepsis. Int J Lab Hematol. 2019 Jun;41(3):392-396. doi: 10.1111/ijlh.12990. Epub 2019 Feb 26. PMID 30806482
- [Background] Soh JS, Lim SW. Delta neutrophil index as a prognostic marker in emergent abdominal surgery. J Clin Lab Anal. 2019 Jul;33(6):e22895. doi: 10.1002/jcla.22895. Epub 2019 Apr 15. PMID 30985959
- [Background] Jha P, Espinoza N, Webb E, Kohli M, Poder L, Morgan T. Single institutional experience with initial ultrasound followed by computed tomography or magnetic resonance imaging for acute appendicitis in adults. Abdom Radiol (NY). 2019 Jul;44(7):2357-2365. doi: 10.1007/s00261-019-01998-1. PMID 30949783
- [Background] Kim HY, Park JH, Lee SS, Lee WJ, Ko Y, Andersson RE, Lee KH. CT in Differentiating Complicated From Uncomplicated Appendicitis: Presence of Any of 10 CT Features Versus Radiologists' Gestalt Assessment. AJR Am J Roentgenol. 2019 Nov;213(5):W218-W227. doi: 10.2214/AJR.19.21331. Epub 2019 Aug 15. PMID 31414891
- [Background] Rawolle T, Reismann M, Minderjahn MI, Bassir C, Hauptmann K, Rothe K, Reismann J. Sonographic differentiation of complicated from uncomplicated appendicitis. Br J Radiol. 2019 Jul;92(1099):20190102. doi: 10.1259/bjr.20190102. Epub 2019 May 29. PMID 31112397
- [Background] Xu Y, Jeffrey RB, Chang ST, DiMaio MA, Olcott EW. Sonographic Differentiation of Complicated From Uncomplicated Appendicitis: Implications for Antibiotics-First Therapy. J Ultrasound Med. 2017 Feb;36(2):269-277. doi: 10.7863/ultra.16.03109. Epub 2016 Dec 31. PMID 28039865